CLINICAL TRIAL: NCT06088251
Title: Evaluation of Nutrition Training Augmented With Digital Technology in Graduate Medical Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 00005155
Record Dates: First submitted 2023-10-11; First posted 2023-10-18 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Chronic Disease
Keywords: Medical Education; Nutrition Counseling; Technology
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutri Training (Experimental): Nutri Training will begin with 1) a presentation of diet counseling evidence and best practices for advising patients, along with information about nutrition recommendations for patients with chronic illness and 2) tools supporting the patient for follow-up. This content will be delivered via a live demonstration of the Nutri interactive software and case demonstration, a novel approach to delivering the learning objectives of standard nutrition education for residents.
  Interventions: Behavioral: Nutri Training
- Standard Nutrition Education (Active Comparator): Standard Nutrition Training will present an overview of 1) nutrition recommendations for patients with chronic disease and 2) cover the role of a registered dietitian and referrals.
  Interventions: Behavioral: Standard Nutrition Education

INTERVENTIONS:
Behavioral: Nutri Training — Nutri Training will begin with 1) a presentation of diet counseling evidence and best practices for advising patients, along with information about nutrition recommendations for patients with chronic illness and 2) tools supporting the patient for follow-up. This content will be delivered via a live demonstration of the Nutri interactive software and case demonstration, a novel approach to delivering the learning objectives of standard nutrition education for residents.
  Arms: Nutri Training
Behavioral: Standard Nutrition Education — Standard Nutrition Education Standard Nutrition Training will present an overview of 1) nutrition recommendations for patients with chronic disease and 2) cover the role of a registered dietitian and referrals.
  Arms: Standard Nutrition Education

SUMMARY:
Investigators will conduct a randomized controlled evaluation of standard nutrition education vs. standard education + Nutri, and interactive clinical software that automates diet assessment and guides resident physicians through personalized and evidence-based diet counseling. Investigators will evaluate differences in resident-reported diet counseling competence and self-efficacy using survey measures. Investigators will evaluate skills using a simulated patient appointment and coding scheme described in prior work.

ELIGIBILITY:
Inclusion Criteria:

* Dell Medical School Internal Medicine Residents
* Dell Medical School Family Medicine Residents

Exclusion Criteria:

* N/A

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2023-10-24 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Diet Counseling Competence | Resident pre-assessment and post-assessment, expected to be 2 weeks after enrollment
  Self-report of diet counseling competency; 4-point Likert-like scale scale; higher score means better outcome
Diet Counseling Self-Efficacy | Resident pre-assessment and post-assessment, expected to be 2 weeks after enrollment
  Self-report of confidence (self-efficacy) in diet counseling; 4-point Likert-like scale scale; higher score means a better outcome.
Diet Counseling Skills | Post-hoc analysis of simulation activity, expected to be at 2 weeks after training intervention
  We will also use an observation checklist to systematically capture resident shared decision-making and diet counseling skills. We will create this checklist based on a literature review of similar tools, such as the Shared Decision Making (SDM) SDM-9 and the coding scheme described in Alexander 2011. Higher score indicates a better outcome. Score range will be reported once the scale has been finalized.

OTHER OUTCOMES:
Physician Diet Counseling Outcome Expectations | Resident pre-assessment and post-assessment, expected to be 2 weeks after enrollment
  Self-report of diet counseling outcome expectations; 5-point Likert-like scale; higher score means better outcome.
Semi-structured debrief interview | Post-hoc analysis of simulation activity, expected to be at 2 weeks after training intervention
  Semi-structured debrief interview to better understand the resident's experience and feedback on the training session and simulation activity.
Training Satisfaction | Resident post-assessment, expected to be 2 weeks after enrollment
  Self-report of satisfaction with training; 5-point Likert-like scale scale; higher score means a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Marissa Burgermaster, PhD, Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin - Burgermaster Lab, Austin, Texas, United States

REFERENCES:
- [Background] Alexander SC, Cox ME, Boling Turer CL, Lyna P, Ostbye T, Tulsky JA, Dolor RJ, Pollak KI. Do the five A's work when physicians counsel about weight loss? Fam Med. 2011 Mar;43(3):179-84. PMID 21380950
- [Background] Jay M, Gillespie C, Ark T, Richter R, McMacken M, Zabar S, Paik S, Messito MJ, Lee J, Kalet A. Do internists, pediatricians, and psychiatrists feel competent in obesity care?: using a needs assessment to drive curriculum design. J Gen Intern Med. 2008 Jul;23(7):1066-70. doi: 10.1007/s11606-008-0519-y. PMID 18612746
- [Background] Kriston L, Scholl I, Holzel L, Simon D, Loh A, Harter M. The 9-item Shared Decision Making Questionnaire (SDM-Q-9). Development and psychometric properties in a primary care sample. Patient Educ Couns. 2010 Jul;80(1):94-9. doi: 10.1016/j.pec.2009.09.034. Epub 2009 Oct 30. PMID 19879711
- [Background] Vetter ML, Herring SJ, Sood M, Shah NR, Kalet AL. What do resident physicians know about nutrition? An evaluation of attitudes, self-perceived proficiency and knowledge. J Am Coll Nutr. 2008 Apr;27(2):287-98. doi: 10.1080/07315724.2008.10719702. PMID 18689561